CLINICAL TRIAL: NCT03397862
Title: A Randomized Double-Blind Study to Assess the Skin Irritation and Sensitization Potential of Once-Weekly Corplex™ Donepezil Transdermal Delivery System
Brief Title: A Skin Irritation Assessment of Once-Weekly Corplex™ Donepezil Transdermal Delivery System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corium, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: P-16011
Record Dates: First submitted 2017-11-03; First posted 2018-01-12 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Skin Irritation; Sensitization

STUDY DESIGN:
Intervention Model Description: Induction Phase will consist of application of the once-weekly TDS for 3 consecutive weeks to the same skin site, followed by a rest period of 2 weeks. The TDS application site will be visually scored for skin irritation approximately 30 minutes following each patch removal and prior to the next patch application. The Challenge Phase will consist of 2 days of TDS application followed by 3 days of visual scoring of TDS application site following TDS removal. Subjects meeting the guidance criteria for Re-Challenge phase will continue with a rest period of 4-8 weeks, followed by 2-day TDS application and a 3-day visual scoring of the TDS application site following TDS removal.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will occur at package level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Corplex Donepezil TDS 5 mg/day (Experimental): Subjects will receive Corplex Donepezil TDS 5 mg/day during Induction, Challenge, and Re-Challenge phase.
  Interventions: Drug: Donepezil TDS
- Vehicle TDS (Placebo Comparator): Subjects will receive Vehicle TDS during Induction, Challenge, and Re-Challenge phase.
  Interventions: Drug: Vehicle TDS

INTERVENTIONS:
Drug: Donepezil TDS — Donepezil patch
  Arms: Corplex Donepezil TDS 5 mg/day
Drug: Vehicle TDS — Placebo patch
  Arms: Vehicle TDS

SUMMARY:
A study to assess the skin irritation and sensitization potential of Corplex™ Donepezil Transdermal Delivery System (TDS)

DETAILED DESCRIPTION:
This study is a multiple center, randomized, double-blind, vehicle-controlled, and multiple-dose study to assess skin irritation and skin sensitization in healthy subjects.

Subjects will be randomized prior to the first TDS application. The total duration of the study from Screening to Follow-up is approximately 95 days for subjects participating in the Induction Phase and the Challenge Phase of the study and potentially up to 156 days for subjects requiring to complete Re-Challenge Phase.

Skin irritation will be monitored by visual scoring scales. TDS adhesion will be assessed during TDS wear period. Safety will be monitored throughout the study by clinical and laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female
* Body mass index ≥ 18.0 and ≤ 35.0 kg/m2
* Medically healthy, as deemed by the Investigator
* Have a skin type with Fitzpatrick scale score of I, II, or III

Exclusion Criteria:

* History or presence of alcoholism or drug abuse
* History or presence of hypersensitivity or idiosyncratic reaction to the study product or related compounds
* Positive urine drug or alcohol results
* Female subjects with a positive pregnancy test or who are lactating
* Any of the following drugs, but not limited to, for 30 days prior to the first dose of study product treatment on Day 1 and throughout the study:

  1. Inducers of cytochrome enzymes and/or P-glycoprotein
  2. Anti-inflammatory drugs or cyclooxygenase 2 analgesics
  3. Beta-blockers
  4. Cholinergics and anticholinergics
  5. Muscle relaxants, anti-Parkinsonian, or neuroleptic medications
* History or presence of significant skin damage deemed by the investigator to potentially interfere
* Any medical or surgical procedure or trauma
* Participation in another clinical study within 30 days or 5 times the half-life of the investigational product (whichever is longer) prior to the first study product treatment

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Mean Cumulative Skin Irritation Score of Donepezil Corplex TDS (Induction Phase) | Induction (21 days)
  Mean Cumulative skin irritation score is determined by averaging the combined Dermal Response score (8-point categorical scale using numeric values) and the Other Effects score (6-point categorical scale using alphabet letters equivalent to numeric values) during the induction phase of the study.
Number of Subjects with Skin sensitization potential of Corplex TDS (Challenge Phase) | Challenge: Up to 5 days including 2-day TDS application and a 3-day visual scoring of the TDS application site following TDS removal
  Subject's sensitization potential will be assessed using the combined Dermal Response score (8-point categorical scale using numeric values) and the Other Effects score (6-point categorical scale using alphabet letters equivalent to numeric values) . The last of 48 hr or 72 hr score collected after TDS removal during the Challenge Phase will be assessed. Provided the combined score is 2 or greater, it will then be compared to the skin irritation scores collected during the induction phase. If the last Challenge Phase score is 2 or greater and generally exceeds the skin irritation scores collected during the induction phase, the subject will return for the Re-Challenge phase.
Number of Subjects with Skin sensitization potential of Corplex TDS (Re-Challenge Phase) | Re-Challenge: Up to 5 days including 2-day TDS application and a 3-day visual scoring of the TDS application site following TDS removal
  Subject's sensitization potential will be assessed using the combined Dermal Response score (8-point categorical scale using numeric values) and the Other Effects score (6-point categorical scale using alphabet letters equivalent to numeric values). The last of 48 hr or 72 hr score collected after TDS removal during the Re-Challenge phase will be assessed. The subject will be considered for potential sensitization if they meet the same criteria in both Challenge phase and Re-Challenge phase (i.e. a combined score of 2 or greater at the last assessment at 48 hr or 72 hr post patch removal and the score are generally higher compared to induction phase scores.

SECONDARY OUTCOMES:
Mean Cumulative Skin Irritation Score of Donepezil Corplex TDS compared to Vehicle TDS (Induction Phase) | Induction (21 days)
  Mean cumulative skin irritation will be determined and compared between Corplex Donepezil TDS and Vehicle TDS. Mean Cumulative skin irritation score is determined by averaging the combined Dermal Response score (8-point categorical scale using numeric values) and the Other Effects score (6-point categorical scale using alphabet letters equivalent to numeric values) during the induction phase of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, MD, CPI, Principal Investigator — Celerion; Laura Sterling, MD, MPH, Principal Investigator — Celerion; Vaeling Miller, Study Director — Corium International
Locations (2):
- United States (2):
  - Celerion Inc., Phoenix, Arizona
  - Celerion Inc., Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: No
No plans